CLINICAL TRIAL: NCT00343421
Title: Immunogenicity and Safety of PEDIACEL®, a Combined Diphtheria, Tetanus, Five Component Acellular Pertussis, Inactivated Poliomyelitis and Haemophilus Influenzae Type b Conjugate Vaccine (Adsorbed), Compared to Infanrix®-IPV+Hib When Both Vaccines Are Co-Administered With Prevenar® to Infants and Toddlers at 2, 3, 4 and 12-18 Months of Age
Brief Title: Study to Compare Pediacel® to Infanrix®-IPV+Hib When Both Are Co-Administered With Prevenar® in Infants and Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A5I16
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis; Haemophilus Influenzae Type b
Keywords: Diphtheria; Tetanus; Pertussis; Poliomyelitis; Haemophilus influenzae type b; Pneumococcal infections
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Haemophilus Infections; Pneumococcal Infections | interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; Heptavalent Pneumococcal Conjugate Vaccine; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): PEDIACEL co-administered with Prevenar
  Interventions: Biological: PEDIACEL® and Prevenar®
- Group 2 (Active Comparator): Infanrix-IPV+Hib co-administered with Prevenar
  Interventions: Biological: Infanrix®-IPV+Hib and Prevenar®

INTERVENTIONS:
Biological: PEDIACEL® and Prevenar® — 0.5 mL each, IM (opposite thigh)
  Other Names: PEDIACEL®: DT5aP-IPV-Hib 5-component Pertussis vaccine; Prevenar®: Pneumococcal saccharide conj. vaccine, adsorbed
  Arms: Group 1
Biological: Infanrix®-IPV+Hib and Prevenar® — 0.5 mL each, IM (opposite thigh)
  Other Names: Infanrix®-IPV+Hib: DTap, IPV and adsorbed conjugated Hib; Prevenar®: Pneumococcal saccharide conj vaccine, adsorbed.
  Arms: Group 2

SUMMARY:
The purpose of this study is to evaluate safety and immunogenicity of Pediacel® in infants and toddlers when given at 2,3,4 and 12-18 months of age.

Primary Objectives:

* To compare the post-dose 3 immunogenicity of Pediacel® to Infanrix®-IPV+Hib when both are co-administered with Prevenar®.
* To describe the post-dose 3 pertussis antibody responses.

Secondary Objectives:

* To compare the post-dose 4 immunogenicity of Pediacel® to Infanrix®-IPV+Hib when both are co-administered with Prevenar®.
* To describe the safety after each vaccination following co-administration with Prevenar®.

ELIGIBILITY:
Inclusion Criteria:

* Infants 55 to 75 days old, inclusive on the day of first vaccination
* Born at full term of pregnancy (> 37 weeks)
* Informed consent form signed by the parent(s) or the legal guardian
* Parents or the legal guardian able to read and write in the local language
* Parent(s) or the legal guardian able to attend all scheduled visits and to comply with the study procedures.

Exclusion Criteria:

* Presence of fever (defined as rectal body temperature ≥ 38.0°C) reported within the last 72 hours
* Moderate or severe acute illness with or without fever
* Participation in another clinical trial in the 30 days preceding first study vaccination
* Planned participation in another clinical trial during the present study period
* Received diphtheria, tetanus, pertussis, poliomyelitis, Haemophilus influenzae type b or a pneumococcal vaccine separately or in combination prior to study vaccination
* Received any vaccination in the 30 days preceding the first study vaccination and/or is planning any vaccination within 6 weeks following any of the study vaccinations
* Congenital or acquired humoral/cellular immunodeficiency or immunosuppressive therapy such as long-term systemic corticosteroids therapy (≥ 2 mg/kg/day prednisone equivalent for ≥ 14 days) in the previous 30 days
* Systemic or local hypersensitivity to any of the study vaccine components (including neomycin, streptomycin, polymyxin B and formaldehyde)
* History of life-threatening reaction(s) (such as encephalopathy, Hypotonic-Hyporesponsive Episode, rectal body temperature ≥ 40.0°C, convulsions with or without fever) to any vaccine containing the same components as the study vaccines
* Blood or blood-derived products (immunoglobulins) received since birth
* Known Human immunodeficiency virus (HIV) seropositivity
* Known thrombocytopenia or other bleeding disorder contraindicating intramuscular vaccination
* History of encephalopathy, seizures or progressive, evolving or unstable neurological condition
* Clinically significant findings on review of systems that might interfere with study vaccination or which, in the opinion of the Investigator, would interfere with the evaluation of the study vaccine/objectives or pose a health risk to the subject.

Ages: 55 Days to 75 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 588 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of PEDIACEL® and Infanrix®-IPV+Hib | 1 month post-vaccination

SECONDARY OUTCOMES:
To provide information concerning the safety after administration of PEDIACEL® and Infanrix®-IPV+Hib | Entire study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Paris, France
- Poznan, Poland

REFERENCES:
- [Result] Grimprel E, Wysocki J, Boisnard F, Thomas S, Mwawasi G, Reynolds D. Immunogenicity and safety of fully liquid DTaP(5)-IPV-Hib compared with DTaP(3)-IPV/Hib when both coadministered with a heptavalent pneumococcal conjugate vaccine (PCV7) at 2, 3, 4, and 12 to 18 months of age: a phase III, single-blind, randomised, controlled, multicentre study. Vaccine. 2011 Oct 6;29(43):7370-8. doi: 10.1016/j.vaccine.2011.07.078. Epub 2011 Jul 30. PMID 21807056
- See also: Related Info — http://www.sanofipasteur.com